CLINICAL TRIAL: NCT03563105
Title: Assessment of Circulatory Compromise With Ox-Imager Using a Vascular Occlusion Test Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Modulated Imaging Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 900-0003
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Circulatory; Change
Keywords: tissue oxygen saturation

STUDY DESIGN:
Intervention Model Description: Vascular Occlusion Test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Desaturation (Experimental): Vascular Occlusion Test
  Interventions: Device: The Ox-Imager Mini (Desaturation)

INTERVENTIONS:
Device: The Ox-Imager Mini (Desaturation) — Vascular Occlusion Test

SUMMARY:
The objective of this study is to evaluate the performance of Modulated Imaging Inc.'s (MI) next generation Spatial Frequency Domain Imaging (SFDI) system to measure potential circulatory compromise.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the performance of Modulated Imaging Inc.'s (MI) next generation Spatial Frequency Domain Imaging (SFDI) system, "The Ox-Imager Mini". Potential circulatory compromise will be imaged in healthy volunteers using both the subject and predicate devices (Ox-Imager CS) in a Vascular Occlusion Test (VOT) model. The VOT model is an established paradigm to introduce transient ischemia in skin and the the subjects will be imaged during this time. The primary endpoint will be to measure significant decrease in tissue oxygen saturation after occlusion for both predicate and subject devices.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age

Exclusion Criteria:

* History of congestive heart failure
* Patients with existing wound or ulcer.
* Rheumatoid arthritis
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Significant decrease in StO2 during occlusion | immediate
  significant decrease in StO2 during occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Amaan Mazhar, PhD, Principal Investigator — Modulated Imaging Inc.
Locations (1):
- Orange County Wound and Hyperbaric, Santa Ana, California, United States